CLINICAL TRIAL: NCT00475605
Title: APPLES: A Prospective Pediatric Longitudinal Evaluation to Assess the Long-Term Safety of Tacrolimus Ointment for the Treatment of Atopic Dermatitis
Brief Title: A Pediatric Longitudinal Evaluation to Assess the Long-Term Safety of Protopic for the Treatment of Atopic Dermatitis
Acronym: APPLES
Status: Terminated | Type: Observational
Why Stopped: Terminated early, endorsed by the FDA based on futility of continuation.
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: F506-CL-5801; FG506-06-37 (Other: Sponsor); 03-0-161 (Other: Sponsor (Astellas)); EUPAS (Registry Identifier: EUPAS12360); LP0156-1294 (Other: Sponsor (LEO Pharma A/S))
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; child; tacrolimus ointment; Protopic Ointment
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1. Protopic Exposure: Pediatric subjects whose ages are/were <16 years at the time of first tacrolimus ointment exposure

SUMMARY:
This is an observational study to assess the long-term safety of Protopic® Ointment for the treatment of atopic dermatitis. Patients whose ages are/were < 16 years at the time of first tacrolimus ointment exposure are eligible to participate. No drug is distributed during this observational trial.

DETAILED DESCRIPTION:
Data will be collected at enrollment and every 6 months thereafter either by interview, Internet, or physician office visit. Each subject will be followed for 10 years in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who first used Protopic® 0.03% or 0.1% before they were sixteen years of age and were treated for at least 6 weeks for the treatment of Atopic dermatitis may enroll into the study.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects whose ages are/were <16 years at the time of first tacrolimus ointment exposure
Sampling Method: Non-Probability Sample
Enrollment: 8071 (Actual)
Dates: Start 2005-05-25 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of systemic or cutaneous malignancy | 10 years
  Standardised Incidence Ratio (versus population cancer rates)

CONTACTS AND LOCATIONS:
Overall Officials: LEO Pharma A/S, Study Director — Medical Expert
Locations (311):
- United States (198):
  - Shelby Dermatology, Alabaster, Alabama
  - Pediatric Care Center of NE Alabama, Anniston, Alabama
  - Total Skin and Beauty Dermatology Center, Birmingham, Alabama
  - Metro Pediatrics, P.C, Birmingham, Alabama
  - Pediatric & Adult Asthma and Allergy, P.C., Birmingham, Alabama
  - Skin Wellness Center of Alabama, Birmingham, Alabama
  - Southview Dermatology, Birmingham, Alabama
  - Ruth A Yates, Huntsville, Alabama
  - Alliance Dermatology, Phoenix, Arizona
  - Derma, Phoenix, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Hull Dermatology, P.A., Rogers, Arkansas
  - Coastal Allergy Care, Camarillo, California
  - Tien Nguyen, Fountain Valley, California
  - Dermatology Research Associates, Los Angeles, California
  - California Skin Institute, Mountain View, California
  - Capital Allergy & Respiratory Disease Center, Roseville, California
  - Allergy and Immunology Clinic, San Diego, California
  - Rady Children's Hospital San Diego, San Diego, California
  - California Dermatology Care, San Ramon, California
  - Connecticut Children's Medical Center Dept of Dermatology, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Webster Dermatology, PA, Hockessin, Delaware
  - Atlantic Skin & Cosmetic Surgery Group, Wilmington, Delaware
  - Center for Dermatology, Boca Raton, Florida
  - Angelos Koutsonikolis, MD, PA, Boynton Beach, Florida
  - Joshua Berlin P.A., Boynton Beach, Florida
  - Fort Lauderdale Dermatology & Cosmetic Skin Center, Fort Lauderdale, Florida
  - North Florida Dermatology Associates, P.A., Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Andrea Trowers, MD, North Miami, Florida
  - Tory Patrick Sullivan, North Miami Beach, Florida
  - Allergy Associates of the Palm Beaches, PA, North Palm Beach, Florida
  - Orlando Dermatology, Orlando, Florida
  - Donna Zeide, Palm Beach Gardens, Florida
  - Waterman Dermatology, Plantation, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Dr.Robert A. Norman, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc, Albany, Georgia
  - Emory University, Atlanta, Georgia
  - Dermatology Consultants PC, Covington, Georgia
  - Dermatologic Surgery Specialist Inc., Macon, Georgia
  - MedaPhase,Inc., Newnan, Georgia
  - AeroAllergy Research Labs of Savannah, Inc., Savannah, Georgia
  - Southern Crescent Dermatology, Stockbridge, Georgia
  - Paul S. Takiguchi- MD- Inc., ‘Aiea, Hawaii
  - Wayne Fujita, M.D. - Private Practice, ‘Aiea, Hawaii
  - Dermatology Clinic of Idaho, Boise, Idaho
  - Southeast Idaho Family Practice, Idaho Falls, Idaho
  - DermAssociates LTD, Belleville, Illinois
  - Christie Clinic, Champaign, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Dermatology, Inc., Carmel, Indiana
  - Shideler Clinical Research Center, Carmel, Indiana
  - Dermatology Associates, PC, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Dermatology Center, New Albany, Indiana
  - Dermatology Center of Indiana P.C., Plainfield, Indiana
  - Randall Dermatology, West Lafayette, Indiana
  - Clinton Urgent Care, Clinton, Iowa
  - Midwest Dermatology, Overland Park, Kansas
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Kansas Medical Clinic, PA, Topeka, Kansas
  - Mid-Kansas Dermatology Clinic, PA, Wichita, Kansas
  - Melissa Knuckles, Corbin, Kentucky
  - Michael W. Simon, M.D., Nicholasville, Kentucky
  - LA Dermatology Assoc LLC, Baton Rouge, Louisiana
  - Kids First Prytania, New Orleans, Louisiana
  - All Kids Pediatrics of Opelousas APMC, Opelousas, Louisiana
  - Holliway Pediatric Clinic, Shreveport, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - Wee Care Pediatrics & Kidmed Clinic, Shreveport, Louisiana
  - Healing Hands Family Medicine, Shreveport, Louisiana
  - Dimitri Dermatology, Slidell, Louisiana
  - Johns Hopkins University, Division of Pediatric Dermatolgy, Baltimore, Maryland
  - Clarksburg Pediatrics, LLC, Clarksburg, Maryland
  - Family Allergy & Asthma Care, Gaithersburg, Maryland
  - Callender Skin and Laser Center, Glenn Dale, Maryland
  - DermAssociates, PC, Silver Spring, Maryland
  - Beverly Johnson, MD, Silver Spring, Maryland
  - Robert S. Berger, White Plains, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Adult & Pediatric Dermatology, Marlborough, Massachusetts
  - Kenneth M. Reed, MD, Quincy, Massachusetts
  - Drs. Iacobelli & DiGregorio, PC, Clinton Township, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Silverton Skin Institute, Grand Blanc, Michigan
  - SVC Dermatology PC, Sterling Heights, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Grekin Skin Institute, Warren, Michigan
  - Midwest Center for Dermatology and Cosmetic Surgery, Warren, Michigan
  - Dermatology Center for Children and Young Adults, Eagan, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Asthma & Allergy Center of North Jackson, Jackson, Mississippi
  - Peace Children's Clinic, Jackson, Mississippi
  - North County Dermatology, Florissant, Missouri
  - Kosse Pediatrics, Saint Joseph, Missouri
  - South Lincoln Dermatology Clinic, Lincoln, Nebraska
  - Skin Specialists PC, Omaha, Nebraska
  - Bettencourt Skin Center, Henderson, Nevada
  - Aistheta, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cheryl D. Ackerman, Glen Ridge, New Jersey
  - CDLC, Ridgewood, New Jersey
  - The Dermatology Group, PC, Verona, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Allergy & Asthma Associates of NNM, Los Alamos, New Mexico
  - New York Dermatology, P.C., Bayside, New York
  - Robert S. Darr, MD, PC, Brooklyn, New York
  - Morris Westfried, M.D., Brooklyn, New York
  - Garden City Dermatology, P.C., Garden City, New York
  - Hollis Medisys, Hollis, New York
  - Marvin S.Watsky, Lindenhurst, New York
  - Orange Dermatology Assoc, PC, Monroe, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Columbia University Medical Center., Dept. of Medicine, New York, New York
  - Helendale Dermatology & Medical Spa, LLC, Rochester, New York
  - Marina I Peredo, MD, Smithtown, New York
  - Derm Research Center of New York, Inc., Stony Brook, New York
  - Joseph D. Sutton, MD, Suffern, New York
  - Stanley A. Newfield, Valley Stream, New York
  - Davie Dermatology, Advance, North Carolina
  - Alamance Skin Center, Burlington, North Carolina
  - Pediatrx Clinic, Fayetteville, North Carolina
  - Southeastern Dermatology, PA, Lumberton, North Carolina
  - FMC/OIC, Rocky Mount, North Carolina
  - DermOne Dermatology Center, PA, Wilmington, North Carolina
  - Carolina Dermatology & Skin Cancer Surgery, Wilmington, North Carolina
  - Knox Clinic Pediatrics, PLLC, Wilmington, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Haber Dermatology and Cosmetic Surgery, Inc, Beachwood, Ohio
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - Dermatology Research Associates, Inc., Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Warren Dermatology & Allergy, Warren, Ohio
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Brian Lepley, D.O., Oklahoma City, Oklahoma
  - Family Health Center South, Oklahoma City, Oklahoma
  - OSU-CHS Houston Center Physicians, Tulsa, Oklahoma
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - East Penn Dermatology, North Wales, Pennsylvania
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - Cheraw Pediatrics, P.A., Cheraw, South Carolina
  - Dermatology Group LLC, Columbia, South Carolina
  - McClerklin Skin and Laser Center, Columbia, South Carolina
  - Allergic Disease & Asthma Center, Greenville, South Carolina
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Palmetto Skin & Laser Center, Rock Hill, South Carolina
  - The Asthma Institute PLLC, Chattanooga, Tennessee
  - Rivergate Dermatology Research Center, Goodlettsville, Tennessee
  - Dermatology Associates of Kingsport, PC, Kingsport, Tennessee
  - Allergy Associates, PA dba East Tennessee Center for Clinical Research, Knoxville, Tennessee
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - The Skin Wellness Center, Knoxville, Tennessee
  - Sheffield Pediatrics, PLLC, Memphis, Tennessee
  - Raleigh Group PC, Memphis, Tennessee
  - Academy of Clinical Research, Arlington, Texas
  - Arlington Center for Dermatology, Arlington, Texas
  - Zoltan Trizna, Austin, Texas
  - Allergy Partners North Texas Research, Dallas, Texas
  - Dermatology Treatment and Research Center, PA, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - University of N. Texas Health Science Center, Fort Worth, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Dermatology Center of Frisco, Frisco, Texas
  - Pediatric Dermatology of North Texas PA, Grapevine, Texas
  - Stephen Schwartz, Harlingen, Texas
  - Heights Dermatology & Aesthetic Center, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - West Houston Dermatology, PA, Houston, Texas
  - Bear Creek Clinic, PA, Houston, Texas
  - Lone Star Children's Medical PLLC, Houston, Texas
  - Dermatology and Laser Center, Irving, Texas
  - Site US0048, Irving, Texas
  - Lubbock Dermatology and Skin Cancer Center, Lubbock, Texas
  - Rick Lin, D.O., MPH, McAllen, Texas
  - Pasadena Dermatology Clinic, Pasadena, Texas
  - Medical Research Network, Spring, Texas
  - Dermatology Research Associates of Tyler, Tyler, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Brookside Pediatrics, Bennington, Vermont
  - Glenn H. Fuchs, MD PC, Arlington, Virginia
  - Dermatology Assoc of Northern Vineland, Centreville, Virginia
  - Piedmont Dermatology Center, PC, Martinsville, Virginia
  - Children's Hospital of the Kings Daughters, Norfolk, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, PLLC, Seattle, Washington
  - Asthma, Inc., Seattle, Washington
  - Eastern Washington Dermatology, Walla Walla, Washington
  - Univeristy of Wisconsin-Madison, Madison, Wisconsin
  - George V. Chandy MD SC, Milwaukee, Wisconsin
  - Central Wyoming Skin Clinic, Casper, Wyoming
- Austria (3):
  - LKH Feldkirch, Feldkirch
  - Landesfrauen- und -kinderklinik, Linz
  - Salzburger Landeskliniken, Salzburg
- Canada (7):
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research, Inc., St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Association, Halifax, Nova Scotia
  - Sudbury Skin Clinic, Greater Sudbury, Ontario
  - Mediprobe Research, Inc., London, Ontario
  - Lynderm Research, Inc., Markham, Ontario
- France (24):
  - Cabinet Medical, Amiens
  - Hopital Pellegrin, Bordeaux
  - Cabinet de Dermatologie - Boulogne-Sur-Mer, Boulogne
  - Cabinet de Dermatologie - Boulogne, Boulogne
  - Hopital Augustin Morvan, Brest
  - Cabinet de dermatologie - Cannes, Cannes
  - Hopital Trousseau, Chambray-lès-Tours
  - Polyclinique du Cotentin, Équeurdreville-Hainneville
  - Centre Hospitalier, Le Mans
  - Hopital Claude Huriez, Lille
  - Cabinet de Dermatologie - Martigues, Martigues
  - Hopital de l'Hotel Dieu, Nantes
  - Cabinet Dermatologie, Nantes
  - Cabinet de Dermatologie, Nice
  - Cabinet de Dermatologie - Paris, Paris
  - Hospital Saint Louis, Paris
  - Hospital Necker, Paris
  - CHU La MILETRIE Service de Dermatologie, Poitiers
  - HOPITAL CHARLES NICOLLE Service de Dermatologie, Rouen
  - Hopital Nord, Saint-Priest-en-Jarez
  - Cabinet de Dermatologie-Strasbourg, Strasbourg
  - Cabinet de Dermatologie, Thann
  - Hopital Larrey, Toulouse
  - Centre Hospitalier Service de Dermatologie, Troyes
- Germany (46):
  - Licca Fachklinik f. aesthetisch- operative Dermatologie und Chirurgie, Augsburg
  - Kinderarztpraxis, Bamberg
  - Charite - Universitaetsmedizin Berlin Klinik fuer Dermatologie, Venerologie u. Allergologie, Berlin
  - Hautarztpraxis, Berlin
  - Klinik fuer Kinder u. Jugendmedizin der Ruhr Universitaet Bochum im St.-Josef-Hospital, Bochum
  - Universitaet Bonn Klinik und Poliklinik fuer Dermatologie, Bonn
  - Hautarztpraxis, Bremen
  - Dermatologisches Zentrum Buxtehude, Buxtehude
  - Hautarztpraxis, Crimmitschau
  - Hautarztpraxis, Dessau
  - Hautarztpraxis, Dresden
  - Arztpraxis fuer Hautkrankheiten, Dresden
  - Klinik und Poliklinik f. Dermatologie Universitaetsklinikum Dresden, Dresden
  - Hautklinik, Düsseldorf
  - Heinrich-Heine-Universitaet Hautklinik, Düsseldorf
  - Hautklinik des Universitaetsklinikums Erlangen, Erlangen
  - Falker, Gernot, Hautarztpraxis, Frankenberg
  - Universitaetsklinikum Klinische Forschung, Zentrum d. Dermatologie u. Venerologie, Frankfurt
  - Derma-Study-Center-Friedrichshafen, Friedrichshafen
  - Hautarztpraxis, Gelnhausen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Kath. Kinderkrankenhaus Wilhelmstift, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Brinkmann, Hautarztpraxis, Herborn
  - Hautarztpraxis Sempell, Itzehoe
  - Klinikum der Fr.-Schiller-Universitaet, Jena
  - Universitaet Hautklinik Kiel, Kiel
  - DermaKiel-Hautarztpraxis, Kiel
  - Klinik fuer Dermatologie, Venerologie u. Allergologie, Leipzig
  - Johannes-Gutenberg Universitaet, Mainz
  - Universitaetsklinikum Giessen+ Marburg Dermatolgie und Allergologie, Marburg
  - Praxis Dermatologie, Marburg
  - Hautarztpraxis, Markkleeberg
  - Kinder- und Jugendaertzin, Mönchengladbach
  - Ludwig - Maximilians Universitaet, Klinik u. Poliklinik fuer Dermatologie u. Allergologie, München
  - Universitaetsklinikum Muenster, Klinik & Poliklinik Fuer Hautkrankheiten, Münster
  - Proinnovera GmbH, Münster
  - Facharzt f. Kinder-und Jugendmedizin, Münster
  - Facharzt fuer Kinder-und Jugendmedizin, Ravensburg
  - Hautarztpraxis, Riesa
  - Richter - Fachaerztin fuer Kinder- und Jugendmedizin, Solingen
  - Termeer, Christian, Stuttgart
  - Universitaets-Hautklinik Tuebingen, Tübingen
  - Marienhospital Wesel Kinderklinik/Forschungsinstitut, Wesel
  - Kinderarztpraxis, Wesseling
  - Hautarztpraxis, Wusterwitz
- Ireland (3):
  - South Infirmary, Cork
  - Our Lady's Hospital for Sick Children, Dublin
  - The Park Clinic, Dublin
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum St. Radboud, Nijmegen
- Poland (11):
  - Prywatna Praktyka Lekarska "Alergomed", Bydgoszcz
  - Wojewodzki Szpital Dzieciecy im. J. Brudzinskiego w Bydgoszczy, Wojewodzka Przychodnia Specjalistyczna Dla Dzieci Poradnia ermatologiczna, Budynek "A", Bydgoszcz
  - Private Practice, Bydgoszcz
  - Szpital Dzieciecy Specjalistyczny Z.O.Z. nad Matka i Dzieckiem, Gdansk
  - Praktyka Lekarska, Gostynin
  - SPZOZ Szpital Specjalistyczny im. S. Zeromskiego, Krakow
  - Dermoklinika, Lodz
  - NZOZ Centrum Alergologii, Lodz
  - Alergovita, Lublin
  - Indywidualna Specjalistyczna Praktyka Lekarska, Sierpc
  - NZOZ Przychodnia Dermatologiczna DERMED s.c, Torun
- United Kingdom (16):
  - Amersham Hospital, Department of Dermatology, Amersham
  - Birmingham Children's Hospital, Birmingham
  - Royal Bolton Hospitals Trust, Bolton
  - Addenbrooke's Hospital, Cambridge
  - Wales College of Medicine, Cardiff University, Heath Park, Cardiff
  - Ninewells Hospital and Medical School, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Harrogate & District Foundation NHS Trust Hospital, Harrogate
  - Leeds General Infirmary, Dept of Dermatology, Leeds
  - Site UK3007, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Royal Free Hospital, London
  - Department of Pediatric Allergy and Immunology, Manchester
  - Chase Farm Hospital, Middlesex
  - George Eliot Hospital, Nuneaton
  - University of Manchester, Dermatology-Pharmacology Unit Hope Hospital, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D3T01.1J No increased risk of cancer in children using topical tacrolimus for atopic dermatitis: A 10-year prospective cohort study Prof. Dr. Regina Fölster-Holst - Germany 12 October 2019 11:00 - 11:15 EADV 2019